CLINICAL TRIAL: NCT02293434
Title: Nutritional Status on Admission to Pediatric Intensive Care: A French Multicentric Study
Brief Title: Nutritional Status on Admission to Pediatric Intensive Care
Acronym: NUTRI-REAPED
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9251
Record Dates: First submitted 2014-08-11; First posted 2014-11-18 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Malnutrition; Dwarf - Nutritional
Keywords: Malnutrition; Status Nutritional Weight; Pediatric intensive care
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All Children (1 month to 18 years): All children (1 month to 18 years) admitted to all PICUs in France during three one-week periods (February, June, October) in the course of a year

SUMMARY:
Study rationale: Children admitted to intensive care are often chronically ill and the intensive care setting may upset the balance between nutritional intakes and needs.

As malnutrition is a key factor in the morbidity/mortality on pediatric intensive care units (PICUs), screening for malnutrition and the individualized adaptation of nutritional support are important elements of patient care. Yet no recent study has evaluated the nutritional status of children admitted to PICUs in France.

Primary Objective: Determine the prevalence of malnutrition in the population of children admitted to intensive care.

Secondary objectives:

* Determine the children's nutritional status on admission.
* Characterize the profile of malnourished patients compared with those not malnourished (sex, age, history, chronic disease, usual dietary habits, reason for admission, scheduled/unscheduled admission, surgery/medication, seriousness, seasonality).
* Describe the practices regarding nutritional care in each center.

Population: All children (1 month to 18 years) admitted to all PICUs in France during three one-week periods (February, June, October) in the course of a year.

DETAILED DESCRIPTION:
Study rationale: Children admitted to intensive care are often chronically ill and the intensive care setting may upset the balance between nutritional intakes and needs.

As malnutrition is a key factor in the morbidity/mortality on pediatric intensive care units (PICUs), screening for malnutrition and the individualized adaptation of nutritional support are important elements of patient care. Yet no recent study has evaluated the nutritional status of children admitted to PICUs in France.

Primary Objective: Determine the prevalence of malnutrition in the population of children admitted to intensive care.

Secondary objectives:

* Determine the children's nutritional status on admission.
* Characterize the profile of malnourished patients compared with those not malnourished (sex, age, history, chronic disease, usual dietary habits, reason for admission, scheduled/unscheduled admission, surgery/medication, seriousness, seasonality).
* Describe the practices regarding nutritional care in each center.

Study design:

* Type of study: Observational, descriptive, transversal, and multicentric.
* Population: All children (1 month to 18 years) admitted to all PICUs in France during three one-week periods (February, June, October) in the course of a year.
* Primary assessment parameter: Malnutrition, as defined by the body mass index (BMI) value <-2 SD, according to the WHO Child Growth Standards.
* Factors studied:

  * Nutritional status on admission based on the measurement of simple anthropometric parameters: weight (W), height (H), head circumference (HC) and mid-upper arm circumference (MUAC), which are then used to calculate malnutrition indices.
  * Profile of malnourished patients in relation to hospitalization parameters (age, sex, reason for admission, history, dietary habits).
  * Nutritional practices in PICUs assessed with two questionnaires (medical and nursing) sent to all participating hospitals.
* Sample size: Number of subjects needed to estimate the prevalence of malnutrition, based on the data in the literature with a confidence interval of 95%±3.2%: 600.

ELIGIBILITY:
Inclusion Criteria:

* All children (1 month to 18 years) admitted to all PICUs in France during three one-week periods (February, June, October) in the course of a year.

Exclusion Criteria:

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children (1 month to 18 years) admitted to all PICUs in France
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Nutritional status | Baseline
  Nutritional status (measurement of simple anthropometric parameters, which are then used to calculate malnutrition indices) on admission

SECONDARY OUTCOMES:
Nutritional practice in PICUs | 1 day ( once during the study)
  Nutritional practice in PICUs once during the study : two questionnaires (medical and nursing) sent to all participating hospitals

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien JACQUOT, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France